## ADAPTATION OF COMMUNITY REINFORCEMENT APPROACH FOR THE TREATMENT OF DRUG ADDICTION



**MUHAMMAD SAGHIR** 

DR. MAZHAR IQBAL BHATTI

74-FSS/PHDPSY/F-18

Associate Professor (supervisor)

**Department of Psychology** 

**Faculty of Social Sciences** 

**International Islamic University Islamabad** 

July 10, 2024

## **Consent Form**

I am Muhammad Saghir PhD Scholar, conducting this research under the Department of Psychology at the International Islamic University Islamabad. In this study, experimental research will be carried out using a new treatment approach IICRA (Islamically Integrated Community Reinforcement Approach). All the information obtained will be kept strictly confidential. I kindly request that you voluntarily participate in this research, and you have the full right to withdraw from the study at any stage. Your treatment will be conducted according to this new treatment approach, which is based on the principles of Community Reinforcement Approach (CRA).

| Your signature on this consent form will be required. Thank you for your cooperation | n. |
|---|---|
| Date: | |

Signature: